CLINICAL TRIAL: NCT07182669
Title: Portal Blood Flow and Oxygen Concentration in Subjects With Chronic Mesenteric Ischemia
Brief Title: Blood Flow and Oxygenation in the Portal Vein in Subjects With Chronic Narrowing of the Blood Vessels to the Gut
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulrik Bjoern Andersen, Principal investigator, MD, Consultant, Rigshospitalet, Denmark
Other Study IDs: VEK H-25043058
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Mesenteric Ischemia
Keywords: chronic mesenteric ischemia; fMRI; MRI-TRUST; Portal oxygen concentration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples analyzed for GIP and GLP-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 subjects with mesenteric ischemia: Intake of a meal during the MRI-scan
- 20 subjects with stenosis of mesnteric arteries, but no postprandial pain: Intake of a meal during the MRI-scan

SUMMARY:
In this study the investigators will, with an Magnetic Resonance Imaging (MRI) method, measure the oxygen content in the portal vein, which conduct the blood from the guts to the liver. Examinations will be performed on 20 subjects with meal related abdominal pain due to severe narrowing of the vessels conduction blood to the guts,compared to 20 subjects with similar narrowing of the abdominal vessels, but without meal related pain. The goal of the study is to test a non-invasive, radiation free method to diagnose patients with abdominal pain due to compromized blood supply (chronic mesenteric ischemia).

DETAILED DESCRIPTION:
Chronic mesenteric ischemia is a rare but potentially life threatening disease, in which atherosklerotic narrowing of the blood supply to the guts causes meal related abdominal pain, and subsequent weight loss. While the disease is rare, meal related abdominal pain without narrowing of the vessels to the gut is frequently seen, and, conversely, so is narrowing of the vessels to the gut without pain. This makes the diagnosis difficult. For a clinical diagnosis, meal related pain and weight loss > 5 % of Body Mass Index (BMI) is required together with significant stenosis of the mesenteric vessels. These criteria has the drawback that an unknown number of patients with pain due to ischemia, but not weight loss may exist.

The present study will evaluate the extent of mesenteric ischemia by measuring the oxygen content in the portal vein, using functional MRI with an established technique named T2-Relaxation-Under-Spin-Tagging (TRUST).

Two groups of patients will be examined (20 patients in each group)

1. With a clinical diagnosis of mesenteric ischemia (pain, weight loss, significant stenosis of mesenteric vessels and relief of symptoms after angioplasty.
2. With significant stenosis of the mesenteric vessels, but not meal related pain. The subjects will be examined in a PET-MRI scanner. The flow and oxygen content in the portal vein will be measured in the fasting state and after ingestion of a meal (protein enriched drink). Levels of the gastric peptides GIP, GLP1 and GLP-2 will be evaluated with blood sampling. An injection of 18 F labelled glucose (18F-FDG) will be injected with the purpose of visualising gut sections with reduced uptake due to reduced perfusion with Positron Emission Tomography (PET) scanning.

The primary endpoint will be blood flow and oxygen content in the portal vein, fasting and postprandial, in subjects with mesenteric ischemia defined as improvement of symptoms after angioplasty.

Inclusion criteria:

* Written informed consent
* Male or female persons > 18 years
* Subjects with postprandial abdominal pain considered compatible with mesenteric ischemia, and severe stenosis of the SMA and eventually other mesenteric arteries, diagnosed with CT-angiography or Doppler ultrasound
* OR subjects with severe stenosis of the SMA and eventually other mesenteric arteries, diagnosed with CT-angiography or Doppler ultrasound, but not postprandial pain
* OR subjects with postprandial abdominal pain, but no stenosis of the SMA, verified with Doppler ultrasound.

Exclusion criteria:

* Serious concurrent illness
* BMI > 30
* Cardiac arrhythmia
* Anemia with Hgb < 7,0 mmol/l
* Pregnancy or breastfeeding (urine HCG is performed on all fertile women)
* Systolic blood pressure < 90 or > 200 mmHg
* Claustrophobia
* Patients who, in the judgement of the investigator, is incapable of participating
* Metallic foreign objects in the body, or pacemakers

Design:

Open study with intervention in the form of a standard meal.

Examinations:

Doppler-ultrasound examinations:

The examinations are performed with a GE Logic 10 scanner. Using an abdominal probe, flow in the inferior and superior mesenteric artery and the celiac artery will be examined.

PET- fMRI scans:

All scans will be performed on a Siemens PET-MR scanner.

MR-scans:

Using the scanners body transmit and a four-element SENSE cardiac receive coil, Arterial Spin Labelling (ASL) perfusion and Blood Oxygen Level Dependent imaging (BOLD) T2* will be mapped in the liver. Blood flow will be measured using Phase Contrast Imaging (Q-flow) in the hepatic artery, and the portal vein. Oxygen concentration will be measured using a TRUST sequence in the portal vein and the hepatic vein. All measurements will be performed twice. Some measurements require breath holding for up to 20 seconds.

Analyses:

Blood samples for gastric polypeptides (Glucose Dependent Insulinotrophic Peptide (GIP,) Glucagon Like Peptide 1 (GLP-1), Glucagon Like Peptide 2(GLP-2) and blood glucose ) will be collected after 15 and 30 minutes of supine rest in the fasting state, and after 30 and 60 minutes following the ingestion of the test meal.

Study visits:

There are three study visits:

Day 1: information visit. Before the visit, the patients receive written information and is informed about the possibility of bringing a companion. If the patient is willing to participate, a written declaration of consent is signed.

Day 2: For patients who have not previously had an examination of the mesenteric vessels, a Doppler-ultrasound examination is performed at the department of Clinical Physiology and Nuclear Medicine, Rigshospitalet, Glostrup. The patients meet after an overnight fasting.

Day 3: The patients meet fasting at 8.00 AM at Clinical Physiology and Nuclear Medicine, Rigshospitalet, Blegdamsvej.

The patients meet fasting at 8.00 AM. 250 MBq of 18F-FDG is injected in a cubital vein. They are positioned in the PET-MR-scanner and basal fMRI measurements are performed. Dynamic PET measurements are performed for 40 minutes,followed by a 10 minutes PET-scan. After basal measurements are performed, a standard meal consisting of 2 cans of protein enriched drink is ingested orally. fMRI measurements are continued for 60 minutes.

The duration of the scan will be 90 minutes

Statistical considerations:

Because the minimal relevant difference for portal oxygen concentration is not currently known, a formal power calculation is not possible. As such, this an exploratory study, for which a minimal sample size of sample size of at least 12 per group is recommended. Because significant changes of flow and oxygenation during hand grip exercise and furosemide injection have previously been obtained in a study of 10 normal subjects (11,12), and additionally differences between groups will be assessed, it has pragmatically chosen to include 20 subjects in each group.

Patient discomfort and risks:

For some people, being in an MRI-scanner can be claustrofobic. High noises are emitted during the scan. Otherwise, discomfort or risk of adverse effects are minimal.The scanning will be interrupted immediately in case of any discomfort.

Exposure to ionizing radiation:

The total radiation dose to a patient from 18FFDG is approximately 5 mSv, corresponding to slightly more than the natural background radiation exposure (3 mSv). This is comparable to the radiation dose from a clinical xx scan.

For any mSv, the risk of inducing an incurable cancer disease is theoretically increased by 0,05‰ in addition to the general risk in the population. Thus, a dose of 5 mSv will increase the cancer risk by 0,025% %. This risk is added to the general risk of 25%, which gives a total risk of 25,025 %.

This added risk is considered very small compared to the opportunity to achieve better diagnostic methods that will possibly allow more patients to be correctly diagnosed and treated for the debilitating disease chronic mesenterial ischemia. The MR-methods are even radiation and contrast free.

Ethical considerations:

The study is conducted in accordance with the Helsinki Declaration after approval from the local Scientific Ethical Committee and The Danish Data Protection Agency.

Regardless of the outcome, the results and knowledge obtained from the project is believed to contribute to better and safer investigative methods, and better understanding of the mechanisms behind development and progression of mesenteric ischemia. Hereby, the knowledge obtained may also contribute to a possible improved treatment of these diseases. The investigators believe that potential discomforts and risks are compensated by the expectable advantages of conducting this study.

Participant information/informed consent:

Information on individual data and interpretation hereof will be communicated by the investigator. The participant's right not to know their own data will be respected.

The study is conducted in accordance with the Helsinki Declaration after approval from the local Scientific Ethical Committee and The Danish Data Protection Agency.

No study-specific tests are performed before informed consent for the study is obtained.

Respecting the privacy and physical and mental integrity of the test subjects:

The collection, transfer, storage and analysis of all health-related matters and sensitive personal data including blood samples will be handled according to the data protection act, the general data protection regulation and the law of health.

Financing:

The study was initiated by the responsible physician Ulrik B. Andersen. The Department of Clinical Physiology and Nuclear Medicine, Rigshospitalet, will supply the scans, the tracers and associated goods. The study will otherwise be financed by the investigators. The investigators may seek additional (non commercial) funding.

If funding is received, the ethical committee and the participating patients will be noticed.

ELIGIBILITY:
Inclusion Criteria:

* - Written informed consent
* Male or female persons > 18 years
* Subjects with postprandial abdominal pain considered compatible with mesenteric ischemia, and severe stenosis of the SMA and eventually other mesenteric arteries, diagnosed with CT-angiography or Doppler ultrasound
* OR subjects with severe stenosis of the SMA and eventually other mesenteric arteries, diagnosed with CT-angiography or Doppler ultrasound, but not postprandial pain

Exclusion Criteria:

* - Serious concurrent illness
* BMI > 30
* Cardiac arrhythmia
* Anemia with Hgb < 7,0 mmol/l
* Pregnancy or breastfeeding (urine HCG is performed on all fertile women)
* Systolic blood pressure < 90 or > 200 mmHg
* Claustrophobia
* Patients who, in the judgement of the investigator, is incapable of participating
* Metallic foreign objects in the body, or pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the participating hospital (Copenhagen University Hospital, Rigshospitalet and Copenhagen University Hospital, Hvidovre Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
flow and oxygen concentration in the portal vein | From enrollment Through study completion, an average of 2 years
  Fasting and postprandial flow and oxygen concentration in the portal vein, measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik B Andersen, MD, Consultant, Principal Investigator — Dept. of Clinical Physiology and Nuclear Medicine, Rigshospitalet, Glostrup
Locations (1):
- Dept. of Clinical Physiology and Nuclear Medicine, Copenhagen University Hospital, Rigshospitalet, Copenhagen, State, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication, after motivated request
Supporting Information: CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Forwarded by reasonably motivated request